CLINICAL TRIAL: NCT06695988
Title: Time-restricted Eating Acceptability, Efficacy and Safety in Free-living Adults With Obesity
Brief Title: Time-restricted Eating Acceptability, Efficacy and Safety in Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Responsible Party: Principal Investigator, Nadeeja Wijayatunga, Assistant Professor, University of Mississippi, Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMississippiO
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Time Restricted Eating
Keywords: Time Restricted Eating; Obesity; Intervention; 9 weeks; Randomization; Intermittent fasting
MeSH Terms: conditions — Intermittent Fasting; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating Group (Experimental): The TRE group will consume calorie-containing food and drinks only over an 8-hour window between 6 a.m. to 8 p.m. for 8 weeks. During the fasting period, they can take only calorie-free fluids.
  Interventions: Behavioral: Time Restricted Eating
- Control (No Intervention): They will follow their usual eating patterns and consume food over a period of 12 hours or more.

INTERVENTIONS:
Behavioral: Time Restricted Eating — The intervention group will eat and drink in a prescribed daily feeding window of 8-hour between 6 a.m. to 8 p.m. for 8 weeks and follow their normal exercise and resistance training routines. We will allow +/-1 hour starting and ending times for the eating window while aiming for an 8-hour eating window
  Arms: Time Restricted Eating Group

SUMMARY:
A randomized controlled trial to determine adherence, acceptability and safety of time restricted eating (TRE) in healthy, sedentary, free-living adults with obesity between the ages of 19-65 years when following 16:8 TRE for 8 weeks. This 9-week study includes a baseline week and 8 weeks of the intervention period. Participants are randomly assigned to the TRE or the non-fasting control group. The TRE group will consume calorie containing food and drink only over an 8 hour period and rest of the 16 hour would be fasting. Adherence to TRE and calorie intake are the primary outcomes. Motivators, facilitators and barriers to TRE, hunger and cravings levels, weight bias internalization, body composition (weight, body fat%, fat mass and muscle mass) , Healthy Eating Index (HEI) to assess diet quality, skin carotenoid levels, disordered eating risk, sleep quality, and perceptions of health and well-being are secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 65 years
* Owns a smartphone
* Apparently healthy
* BMI ( more than or equal to 25 kg/m2 ) and high body fat percent (BF%) (≥25% and ≥35% for males and females, respectively)
* Sedentary lifestyle (less than 150 minutes of self-reported moderate to vigorous activity per week)
* Self-reported eating interval of ≥12 h per day

Exclusion Criteria:

* Diagnosed diabetes mellitus (type I or II), coronary heart disease, heart failure, hypertension, hyperlipidemia, stroke, chronic lung diseases, liver or kidney disease, adrenal diseases, musculoskeletal disorders, uncontrolled thyroid disease (dose changes within the past 3 months), Crohn's disease, Ulcerative Colitis, arthritis, undergoing active cancer treatment except for non-melanoma cancer, uncontrolled psychiatric disorder (a history of hospitalization for psychiatric illness).
* Currently taking any medication that is meant for, or has a known effect on, appetite
* On anabolic steroid or hormone replacement therapy
* Participation in an exercise/nutrition/ weight-loss program within the last 6 months
* Any history of surgical intervention for weight management
* Having a ≥5% body weight change during the last 3 months
* Pregnant or less than 6 months post-partum, breastfeeding, polycystic ovarian syndrome or irregular menstruation
* missing limbs, have a pacemaker or metal implants,
* eating disorders or EAT-26 score >20
* Alcohol or drug addiction
* Current smoker
* Works night shifts
* Unable to commit to a 9-week study
* Not willing to follow study protocol and any other contraindications.
* Currently following any of the following restrictive diets - Keto/low carbohydrate/ Vegan/ Vegetarian/ Intermittent fasting/ Paleo/ Calorie restriction/ Any other restrictive diet
* Participating in another study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | 8 weeks
  Percent of days during the 8-week trial when TRE was adhered to as recommended. This will be self-reported daily.
Total calorie intake | During baseline week and week 8 of the intervention
  Pre and post intervention measurements of calorie intake based on three 24-hour food recall surveys using the NDSR software.

SECONDARY OUTCOMES:
Body weight (kg) | At baseline and at the end of 8 weeks of intervention
  Pre and post intervention measures of body weight.
24-hour physical activity energy expenditure (PAEE) | During baseline week and week 8 of the intervention
  GT9X Actigraph accelerometer will be used over 7 days to measure physical activity energy expenditure pre-intervention and during week 8 of the intervention.
Body fat percentage (%) | At baseline and at the end of 8 weeks of intervention
  Pre and post intervention measurements of body fat percentage measured by bioelectrical impedance analyzer.
Fat-free mass (kg) | At baseline and at the end of 8 weeks of intervention
  Pre and post intervention measurements of body fat-free mass (kg) measured by bioelectrical impedance analyzer.
Fat mass (kg) | At baseline and at the end of 8 weeks of intervention
  Pre and post intervention measurements of body fat mass (kg) measured by bioelectrical impedance analyzer.
Hunger and satiety | During baseline week and week 8 of the intervention
  Pre and post intervention subjective measure of hunger and satiety with the use of a Hunger and Satiety Visual Analog Scale
Sleep quality | One time during the baseline week and week 8 of the intervention
  Pre and post intervention measure of subjective sleep quality by use of Pittsburgh Sleep Quality Scale.
Diet Quality | During baseline week and week 8 of the intervention
  Pre and post intervention measurements of diet quality based on three 24-hour food recall surveys at pre- and post collected using the NDSR software and Healthy Eating Index was calculated.
Perceptions of health and well-being | At baseline and at the end of 8 weeks of intervention
  Pre- and post quality of life will be assessed using RAND 36-Item Health Survey 1.0 (SF-36)
Weight Bias Internalization | At baseline and at the end of 8 weeks of intervention
  Pre- and post weight bias internalization will be assessed using the Weight Bias Internalization Scale (WBIS).
Disordered eating risk | At baseline and at the end of 8 weeks of intervention
  Pre- and post disordered eating risk will be assessed using Eating Attitude Test (EAT-26) survey scores
Eating Behavior | At baseline and at the end of 8 weeks of intervention
  Pre and post eating behavior will be assessed using the Three Factor Eating Questionnaire (TFEQ-18). The TFEQ-R18 measures 3 aspects of eating behavior: cognitive restraint, uncontrolled eating, and emotional eating
Skin carotenoid | At baseline and at the end of 8 weeks of intervention
  Pre- and post skin carotenoid levels will be measured pre and post-intervention using a non-invasive NuSkin Biophotonic scanner which is based on the Resonant Raman Spectroscopy technology.
Motivators, barriers, and facilitators for following time restricted eating | At end of 2nd week and during the 8th week of intervention.
  Motivators, barriers, and facilitators when following time restricted eating will be assessed only in the TRE group. These will be collected as qualitative data in the format of a semi-structured interviews over Zoom.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition and Hospitality Management, University of Mississippi, Oxford, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the de-identified participant data used in the published manuscripts by depositing these data in a secure data repository. The data shared will include the sociodemographic data and the outcomes published in the manuscripts. The protocol and statistical analysis plan will be shared as supplementary material through the journal where the study if published, if allowed
Supporting Information: Study Protocol, SAP